CLINICAL TRIAL: NCT05453604
Title: Evaluation Protocols for Isolation of Analytes From Urine for Future Oncology Applications
Acronym: URODETECT-WP1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Novosanis NV (Industry)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019_NOV_CP_001
Record Dates: First submitted 2022-06-24; First posted 2022-07-12 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Prostate Cancer; Urine; Liquid Biopsy
Keywords: Urine; Liquid biopsy; Oncology; Colli-Pee
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sample collection (Experimental): This is a prospective study in which urine samples will be collected from healthy volunteers, urine samples and a blood sample from pregnant women and cancer patients with solid tumors with emphasis on breast- and prostate cancer. The participants will be asked to provide a urine sample collected with the Colli-Pee® device and fill out an online questionnaire to collect usability data.
  Interventions: Device: Colli-Pee UAS devices

INTERVENTIONS:
Device: Colli-Pee UAS devices — Colli-Pee UAS device variants will be evaluated during this study

SUMMARY:
The aim of this study is to evaluate and optimize protocols for the isolation and analysis of analytes in urine (cell-free nucleic acids, extracellular vesicles and proteins). The following factors will be evaluated (1) volumetric collection with Colli-Pee®, a collection device developed by Novosanis for standardized collection of urine, and (2) stabilization methods.

This is a prospective study in which urine samples will be collected from healthy volunteers, urine samples and a blood sample from pregnant women and cancer patients with solid tumors with emphasis on breast- and prostate cancer. The participants will be asked to provide a urine sample collected with the Colli-Pee® device and fill out an online questionnaire to collect usability data. Thereafter, the urine sample will be aliquoted to be used in different pilot studies for the protocol optimization. For the pilot study where the effect of volume will be assessed, participants will be requested to collect multiple samples with different Colli-Pee® variants and fill out questionnaires accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old
* Being able to understand and read Dutch
* For cancer patients specifically: patients suffering from local and systemic cancers (e.g. breast, prostate cancer)

Exclusion Criteria:

* For cancer patients specifically: patients suffering from a blood cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
General DNA or RNA concentration measured using Qubit | Through study completion, an average of 1 year.
  Comparison of DNA or RNA concentrations [ng/µL] measured using Qubit assays
  * between different extraction methods;
  * between different first-void urine volumes (10, 20, 40 mL);
  * between different storage conditions (Day 0, Day 7, Day 14 at room temperature).
Protein concentration measured using ELISA | Through study completion, an average of 1 year.
  Comparison of protein concentrations measured using ELISA assays
  * between different extraction methods;
  * between different first-void urine volumes (10, 20, 40 mL);
  * between different storage conditions (Day 0, Day 7, Day 14 at room temperature).
cell-free DNA or RNA percentages and profiles measured using TapeStation | Through study completion, an average of 1 year
  Comparison of cell-free DNA or RNA percentages (%) and profiles (graphical) measured using TapeStation assays
  * between different extraction methods;
  * between different first-void urine volumes (10, 20, 40 mL);
  * between different storage conditions (Day 0, Day 7, Day 14 at room temperature).
Detection (presence/absence) of specific biomarker targets (SRY, HER2, PIK3CA, AR-V7, TMPRSS2-ERG) for pregnant women, breast cancer patients and prostate cancer patients measured using ddPCR | Through study completion, an average of 1 year
  Comparison of target detection measured using ddPCR assays [copies/µL]
  * between different extraction methods;
  * between different first-void urine volumes (10, 20, 40 mL];
  * between different storage conditions (Day 0, Day 7, Day 14 at room temperature).

SECONDARY OUTCOMES:
Detection (presence/absence) of specific biomarker targets (SRY, HER2, PIK3CA, AR-V7, TMPRSS2-ERG) for pregnant women, breast cancer patients and prostate cancer patients measured using ddPCR. | Through study completion, an average of 1 year
  Comparison of target detection measured using ddPCR assays [positive, negative or copies/µL] in first-void urine samples from all study participants compared to blood testing using ddPCR. (Proof of concept study)
Usability characteristics of the Colli-Pee UAS devices. | Through study completion, an average of 1 year
  All study participants will receive a questionnaire regarding the usability characteristic of the Colli-Pee UAS devices. These questions cover physical information, previous experiences, and usability questions. When scores need to be given participants can score between 0 and 100%, in which 0% is a negative score and 100% is a positive score. When an opinion is asked participants can choose between very difficult, difficult, neutral, easy, and very easy. Analysis will be done using descriptive statistics.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair ziekenhuis Antwerpen, Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No